CLINICAL TRIAL: NCT02725177
Title: Ocular Sarcoidosis Open Label Trial of ACTHAR Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ocular Sarcoidosis 15-1072
Record Dates: First submitted 2016-03-11; First posted 2016-03-31 (Estimated); Results first posted 2023-02-15 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Ocular Sarcoidosis; Panuveitis; Anterior Uveitis
Keywords: Ocular Sarcoidosis
MeSH Terms: conditions — Panuveitis; Uveitis, Anterior | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- H.P. Achtar Gel 80 U (Experimental): H.P. Acthar Gel (repository corticotropin) Injection, 80 U daily for 10 days, then 80 U twice weekly for up to a total of 24 weeks on therapy.
  Interventions: Drug: Repository Corticotropin Injection; Drug: Repository Corticotropin Injection -Treatment Extension

INTERVENTIONS:
Drug: Repository Corticotropin Injection — Treatment with ACTHAR Gel for 24 weeks
  * Initial treatment with 80 units daily for ten days (induction phase)
  * Maintenance treatment with 80 units twice weekly (maintenance phase)
  Other Names: H.P. Acthar Gel; ACTH Gel; ACTH
Drug: Repository Corticotropin Injection -Treatment Extension — 24 open label extension permitted in subjects who respond to treatment
  Other Names: H.P. Acthar Gel; ACTH Gel; ACTH

SUMMARY:
Treatment with ACTHAR Gel will result in a reduction of ocular inflammation in patients with active ocular sarcoidosis that requires systemic immunosuppressant therapy (hypothesis)

DETAILED DESCRIPTION:
The initial treatment of ocular sarcoidosis usually relies on a combination of topical glucocorticoids and oral glucocorticoids, both of which are associated with significant ocular and systemic toxicities. Steroid-sparing therapies are limited by variable and unpredictable efficacy, prolonged time until clinical response, medication intolerance, and difficulties obtaining payor approval. As a result, it is not uncommon that treating physicians must choose between excessive glucocorticoid toxicity versus poor control of ocular inflammation. Ongoing ocular inflammation, in turn, leads to eventual visual loss and occasionally blindness.

There is a need for a more reliable, expeditious therapy that can be used as an alternative to glucocorticoids in sarcoidosis uveitis. Adrenocorticotropic hormone, through activation of melanocortin receptors on leukocytes, can dampen immune responses through non-glucocorticoid dependent mechanisms. The proposed study will aim to define whether there is effectiveness for ACTHAR gel in these patients, delineate an effect dosing regimen, and provide information about the safety of this approach for moderate to severe ocular sarcoidosis.

ACTHAR is a 39-amino acid peptide natural form of adrenocorticotropin hormone (ACTH) that was initially approved in 1952 by the FDA. It has since been approved for 19 indications including respiratory sarcoidosis, multiple sclerosis, and infantile spasms.

ELIGIBILITY:
Inclusion Criteria:

* Patient with sarcoidosis as defined by ATS/ERS/WASOG guidelines (American Thoracic Society/European Respiratory Society /World Association of Sarcoidosis and Other Granulomatous Diseases)
* Any posterior, intermediate or panuveitis of sufficient severity to warrant therapy, in the opinion of the treating physician --OR-- Anterior uveitis requiring 4 or more daily applications of topical corticosteroids to maintain control of inflammation, or uncontrolled with topical therapy
* Persistent disease activity (active uveitis) at the time of screening

Exclusion Criteria:

* Other cause for ocular inflammation
* Uncontrolled diabetes, hypertension, or other contra-indication to increased dosage of glucocorticoids
* Recent (less than 4 weeks) intra-ocular or intra-orbital steroid injection
* Escalation of immunosuppressive medications between screening and initiation of the study medication
* Severe extra-ocular sarcoidosis likely to require additional therapy (in the opinion of the investigator)
* Administration of an investigational medication for sarcoidosis within 3 months, or 5 half-lives, whichever is longer
* Have a history of any opportunistic infection within 6 months prior to screening
* Have any history of malignancy, except fully resected cutaneous squamous cell cancer or cutaneous basal cell cancer, or cervical carcinoma in-situ with a minimum of 5 years period without recurrence
* Severe other organ disease felt to be likely to lead to death within the next six months
* Unable to follow the study protocol, including the requisite travel and follow-up ocular testing
* Women of childbearing potential must be using adequate birth control measures (abstinence, hormonal contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilization) and must agree to continue such precautions, and not become pregnant or plan a pregnancy for 6 months after receiving their last treatment with study agent. Women of childbearing potential must test negative on a serum pregnancy test at screening.
* Breastfeeding women are excluded from participation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Culver, DO, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinical Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- H.P. Achtar Gel 80 U: H.P. Acthar Gel (repository corticotropin) Injection, 80 U daily for 10 days, then 80 U twice weekly for up to a total of 24 weeks on therapy.
  Repository Corticotropin Injection: Treatment with ACTHAR Gel for 24 weeks
  * Initial treatment with 80 units daily for ten days (induction phase)
  * Maintenance treatment with 80 units twice weekly (maintenance phase)
  Repository Corticotropin Injection -Treatment Extension: 24 open label extension permitted in subjects who respond to treatment
Period: Overall Study
Arm/Group | H.P. Achtar Gel 80 U
Started | 9
Completed | 4
Not Completed | 5
Not completed — Physician Decision | 4
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | H.P. Achtar Gel 80 U
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 51 [35 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Clinically Significant Improvement in Visual Acuity
Description: The primary outcome was percentage of patients meeting at least one of the following variables 1) improved visual acuity, 2) resolution of intraocular inflammation, 3) ability to taper ocular or oral steroids by at least 50% or 4) reduction of cystoid macular edema, with no worsening of any single one and no need for additional sarcoidosis therapies at 24 weeks .
Time Frame: Measured at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | H.P. Achtar Gel 80 U
Number analyzed (Participants) | 9
Participants | 3

2. Secondary Outcome: Percentage of Patients With Clinically Significant Improvement in the Resolution-intraocular Inflammation
Time Frame: Measured at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | H.P. Achtar Gel 80 U
Number analyzed (Participants) | 4
Participants | 2

3. Secondary Outcome: Proportion of Patients Experiencing a Tapering of Ocular/Oral Steroids by at Least 50%
Time Frame: Measured at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | H.P. Achtar Gel 80 U
Number analyzed (Participants) | 4
Participants | 2

4. Secondary Outcome: Proportion of Patients With a Clinically Significant Reduction-cystoid Macular Edema
Time Frame: Measured at 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | H.P. Achtar Gel 80 U
Number analyzed (Participants) | 4
Participants | 1

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | H.P. Achtar Gel 80 U
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 7/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | H.P. Achtar Gel 80 U (N=9)
Fluid Retention (Vascular disorders) | 7
Insomnia (General disorders) | 4
Hypertension (Vascular disorders) | 4
Depression (Psychiatric disorders) | 3
Impaired Blood Sugar (Metabolism and nutrition disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT02725177/Prot_SAP_000.pdf